CLINICAL TRIAL: NCT06813027
Title: Use of Allogeneic Extracellular Secretomes (EV)Derived From Umbilical Cord Mesenchymal Stromal Cells: a Phase I Open-label Safety Trial.
Acronym: EVVitiCTC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Jordan (Other)
Collaborators: Abdalla Awidi Abbadi, MD (Unknown)
Responsible Party: Principal Investigator, Hanan Jafar, Principal Investigator, University of Jordan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EV-Vitiliogo-CTC
Record Dates: First submitted 2025-02-03; First posted 2025-02-06 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extracellular vesicles (EV) (Experimental): Extracellular secretomes ( extracellular vesicles "EV") derived from mesenchymal stroma cells (MSCs)
  Interventions: Biological: EV
- Control (No Intervention): No intervention

INTERVENTIONS:
Biological: EV — Extracellular secretomes ( extracellular vesicles "EV") derived from mesenchymal stroma cells (MSCs)
  Arms: Extracellular vesicles (EV)

SUMMARY:
Aim of the study: The primary endpoint of this work is to explore the safety of allogeneic extracellular secretomes "extracellular vesicles" (EV) derived from umbilical cord mesenchymal cells (HUCMSCs) when injected perilesional repeatedly in stable non-facial vitiligo. Methods: Adults with stable non-facial vitiligo for more than three months not exceeding 300 mm 2 were included in the study. A total of 13 patients of either gender, were given perilesional EV weekly for 3 weeks. Adverse events were regularly monitored for six months. The re-pigmentation was assessed at 3 and 6 months The non-injected areas are used as control for comparison of repigmentation. The injected skin area and the control areas were photographed at baseline, at the end of treatment, and at three, and six months.

DETAILED DESCRIPTION:
Vitiligo is an acquired chronic depigmenting disorder of the skin characterized by progressive loss of melanocytes from the epidermis. It clinically manifests as well- demarcated white macules and patches. It affects 0.5%-2% of the global population, irrespective of gender or ethnicity, with significant implications for quality of life (1, 2). The etiology of vitiligo is unknown but is multifactorial, involving genetic, environmental, and immunological factors. Genome-wide association studies have identified over 50 genetic loci associated with the disease, many of which are linked to immune regulation and melanocyte biology (3). Central to its pathogenesis is an autoimmune mechanism, where CD8+ T cells and pro-inflammatory cytokines, such as IFN-γ and TNF-α, mediate melanocyte destruction (4). Oxidative stress and intrinsic melanocyte abnormalities exacerbate immune responses, perpetuating depigmentation. Vitiligo imposes a significant psychosocial burden due to its visible nature. Patients often experience stigmatization, low self-esteem, and anxiety, particularly in cultures where skin appearance is highly valued. Clinically, it is associated with autoimmune comorbidities, including thyroid dysfunction, alopecia areata, and type 1 diabetes, necessitating comprehensive care (5). Therapeutic approaches focus on stopping disease progression and promoting re- pigmentation. Topical steroids and calcineurin inhibitors are first-line treatments for localized disease (6). Narrowband UVB phototherapy remains the gold standard for extensive disease combined with topical agents to improve outcomes (7). Recent advancements in targeted therapies, such as Janus kinase (JAK) inhibitors, have shown promising results in clinical trials, particularly for immune- mediated processes (8). Surgical interventions, including melanocyte transplantation, are viable options for stable disease. Despite these advances, no curative therapy exists, and long-term management remains a challenge. Understanding the interaction of genetic, environmental, and immune mechanisms underlying vitiligo is essential for developing novel, effective treatments. Addressing its psychosocial burden is equally important to improve the quality of life for affected individuals. Extracellular secretomes ( extracellular vesicles "EV") derived from mesenchymal stroma cells (MSCs) have been used in vitiligo in a mouse model. They have been

shown to modulate immune responses, suppress CD8+ T cell-mediated cytotoxicity reduce pro-inflammatory cytokine levels, and promote melanocyte survival (9). In a vitiligo mouse model, EVs from human umbilical cord MSCs were found to cause re-pigmentation by restoring immune homeostasis and protecting melanocytes from apoptosis (9). These findings suggest that EVs could serve as a promising therapeutic tool for vitiligo, providing targeted modulation of immune and melanocyte dynamics in preclinical experiments. No published reports of EV being directly injected into vitiligo-affected areas in humans. This is the first work designed to explore the toxicity and adverse events of an allogeneic EV derived from hucmsc.

ELIGIBILITY:
Inclusion and exclusion criteria Subjects of both genders who were 18 years old or older and had a clinical diagnosis of focal, segmental, or generalized vitiligo that had been stable for more than three months were enrolled.

Additionally, subjects must have normal kidney function, liver function, blood pressure, no heart or lung diseases, and no history of allergies. The following subjects were excluded from the study: those under 18 years of age, pregnant women, patients with new lesions, actively spreading vitiligo, bleeding disorders, active malignancy, heart failure, uncontrolled hypertension, active hepatitis or transmissible disease, history of Koebnerization, history of hypertrophic scars or keloidal tendency, history of allergy, and patients on anticoagulants.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Safety | 6 months
  Safety was the primary endpoint. Adverse events were monitored. Immediately after injection, each subject was kept for one hour of observation in the Cell Therapy Center (CTC). Subjects were followed for 24 hours and then weekly for the first month. Subsequently, they were followed monthly until the end of the study using a special checklist for adverse events as described . Measuring visible adverse events such as redness, localized itching, and skin edema score

SECONDARY OUTCOMES:
Efficacy of response | 6 months
  Efficacy was measured at three and six months. The extent of re-pigmentation was assessed and scored as follows: re-pigmentation of ≤25% Minimal, 26-50% Mild, 51-75% Moderate, 76-90% Marked, and >90% Excellent. All subjects were evaluated clinically using clinical observation and photographs of the affected area at baseline, 3 months, and 6 months. Visual assessment. For each patient, the size (shrinkage or progression of Disease), symptoms (inflammation), and signs (color) were recorded and reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Cell Therapy Center, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No